CLINICAL TRIAL: NCT00610480
Title: Effects of Systane® Versus Optive™ Lubricating Eye Drops in Maintaining Tear Film Stability at Determined Time Points
Brief Title: Tear Film Stability After Instillation of Over-the-Counter (OTC) Artificial Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, V. Vinod Mootha, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 092007-002
Record Dates: First submitted 2008-01-27; First posted 2008-02-08 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Dry Eye Disease
Keywords: Dry Eyes; Tear Film Stability
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optive, then Systane Artificial Tears (Active Comparator): Artificial Tears (Optive, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, artificial tears (Systane, 40 microliters) will be administered using the same procedure protocol.
  Interventions: Drug: 1st visit Optive, then 2nd visit Systane
- Systane, then Optive Artificial Tears (Active Comparator): Artificial Tears (Systane, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, artificial tears (Optive, 40 microliters) will be administered using the same procedure protocol.
  Interventions: Drug: 1st visit Systane, then 2nd visit Optive

INTERVENTIONS:
Drug: 1st visit Optive, then 2nd visit Systane — First visit: Instillation of Optive followed by evaporometry assessment after 30 minutes.
  Second visit: Instillation of Systane followed by evaporometry assessment after 30 minutes.
  Arms: Optive, then Systane Artificial Tears
Drug: 1st visit Systane, then 2nd visit Optive — First visit: Instillation of Systane followed by evaporometry assessment after 30 minutes.
  Second visit: Instillation of Optive followed by evaporometry assessment after 30 minutes.
  Arms: Systane, then Optive Artificial Tears

SUMMARY:
The goal of this research is to evaluate and compare the effectiveness of Systane® versus Optive™ on aqueous tear film stability in patients with a diagnosis of Dry Eye Syndrome and to determine the possible application for this product in the future. Systane® is marketed as over-the-counter tear lubricating therapy in the United States under the FDA monograph.

DETAILED DESCRIPTION:
Twenty (20) patients will be enrolled in this two-period crossover, randomized study design. During the course of the study, each patient will be treated with each test article in the clinic at separate visits. Following the informed consent procedure, a general ocular evaluation, including corneal and conjunctival staining and Schirmer testing, will be done and evaporometry assessments will be completed to determine baseline tear evaporation rate. This will occur before any test article is administered to the patient.

Qualified patients will be randomized into two treatment groups. After 1 hour, in order to eliminate any residual sodium fluorescein, patients will be administered one drop of Systane® (40 µl) or Optive™ (40 µl) in each eye per randomization assignment. At 30 minutes following instillation of the drop, the evaporometry measurement will be repeated. These evaporometry tests (pre and post instillation of drops) will be performed in order to establish a comparison for later analysis. The estimated time in completing each study visit will be 180 minutes per visit. Patients will be asked to return to the clinic after 2 - 14 days for evaluation of the 2nd assigned crossover treatment (i.e. patients who initially received Optive will receive Systane and patients who initially received Systane will receive Optane).

During the interim study periods, patients will be asked to continue their pre-study routine; using their pre-study ocular lubricant or other tear products at the same frequency. Any changes in the frequency of product use during the interim period or any changes in other concomitant medications will be carefully recorded. This is especially important since many prescription products (e.g., Claritan) have significant effects on lacrimal gland physiology.

An effort will be made to schedule all study visits at approximately the same time of day in order to reduce diurnal variability. For the similar reasons, all patients will be asked not to use any lubricants or ocular medications for at least one hour prior to their office visits.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and up will be included, where any age over 89 will be recorded as 'greater than 89.'
* Individuals with bilateral eye sight eye correctable to 20/80 or better.
* Individuals in good health with or without Meibomian Gland Dystrophy (MGD) but with Aqueous Tear Deficiency (ATD) with minimal to no ocular surface inflammation on slit lamp examination.

Exclusion Criteria:

* Individuals with only one sighted eye or vision not correctable to 20/80 or better in both eyes.
* Individuals with history of punctal plugs or punctal occlusions.
* Individuals with history of keratorefractive as well as ophthalmic disease such as corneal dystrophies, glaucoma, or systemic disease affecting the eye (such as Herpes Zoster).
* Individuals with history of systemic or ocular auto-immune conditions.
* Individuals with active systemic disease or those taking systemic medication that are known to influence AT production will not be considered for this trial.
* Individuals using topical medication who are unable to discontinue them for at least 24 hours prior to baseline evaluation will be excluded as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Mootha, MD, Principal Investigator — UTSW Medical Center at Dallas
Locations (1):
- UTSW Medical Center at Dallas - Aston Ambulatory Care Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with dry eye disease will be recruited from Ophthalmology clinic patients and otherwise healthy volunteers who are students or employees of the University of Texas Southwestern Medical Center.
Groups:
- Optive, Then Systane Artificial Tears: Artificial Tears (Optive, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, a baseline evaporation rate will be measured, artificial tears (Systane, 40 microliters) will be administered, and evaporation rate measurements will be repeated 30 minutes later.
- Systane, Then Optane Artificial Tears: Artificial Tears (Systane, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, a baseline evaporation rate will be measured, artificial tears (Optane, 40 microliters) will be administered, and evaporation rate measurements will be repeated 30 minutes later.
Period: Overall Study
Arm/Group | Optive, Then Systane Artificial Tears | Systane, Then Optane Artificial Tears
Started | 10 (10 assigned patients x 2 interventions.) | 10 (10 assigned patients x 2 interventions.)
Completed | 10 (10 assigned patients x 2 interventions.) | 10 (10 assigned patients x 2 interventions.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Optive, Then Systane: Artificial Tears (Optive, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, a baseline evaporation rate will be measured, artificial tears (Systane, 40 microliters) will be administered, and evaporation rate measurements will be repeated 30 minutes later.
- Systane, Then Optive: Artificial Tears (Systane, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, a baseline evaporation rate will be measured, artificial tears (Optane, 40 microliters) will be administered, and evaporation rate measurements will be repeated 30 minutes later.
- Total: Total of all reporting groups
Arm/Group | Optive, Then Systane | Systane, Then Optive | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Aqueous Tear Evaporation Rate Before and After Use of OTC Artificial Tears
Description: To evaluate the effect of OTC artificial tears on tear film stability, the evaporation rate (µl/cm2/min) will be determined with an Evaporometer for the left eye only of each patient. For each arm, the evaporation rates will be determined at baseline and at 30 minutes after installation of artificial tears. Evaporation rates in all cases will be determined under two different relative humidity (RH) conditions, RH from 25-35% and RH from 35-45%.
Time Frame: Baseline and 30 minutes after artificial tear instillation
Population: Total participant enrollment is 20 (3 men and 17 women). Ten participants were assigned to each sequence, so a total of 20 participants experienced each intervention.
Measure: Mean (Standard Deviation); unit: (µl/cm2/min)
Groups:
- Optive Artificial Tears: Artificial Tears (Optive, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, a baseline evaporation rate will be measured, artificial tears (Systane, 40 microliters) will be administered, and evaporation rate measurements will be repeated 30 minutes later.
- Systane Artificial Tears: Artificial Tear
  Artificial Tears (Systane, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later. At the next study visit, 2-14 days later, a baseline evaporation rate will be measured, artificial tears (Optane, 40 microliters) will be administered, and evaporation rate measurements will be repeated 30 minutes later.
Arm/Group | Optive Artificial Tears | Systane Artificial Tears
Number analyzed (Participants) | 20 | 20
(µl/cm2/min)
  Baseline:25-35% | 0.047 (0.019) | 0.049 (0.023)
  Baseline:35-45% | 0.031 (0.014) | 0.032 (0.016)
  30 minutes:25-35% | 0.052 (0.024) | 0.051 (0.025)
  30 minutes:35-45% | 0.034 (0.016) | 0.032 (0.014)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant for up to 2 weeks, from time of enrollment to completion of study visits,
Groups:
- Optive Artificial Tears: Artificial Tears (Optive, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later.
- Systane Artificial Tears: Artificial Tears (Systane, 40 microliters) will be administered at the first study visit, after baseline evaporation rate measurements have been taken. Evaporation rate measurements will be repeated 30 minutes later.
Arm/Group | Optive Artificial Tears | Systane Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes